CLINICAL TRIAL: NCT03098992
Title: Post-market, Prospective, Randomised, Sham-controlled Clinical Trial Designed to Confirm the Efficacy and Safety of the Fotona Smooth® Device to Treat Female Stress Urinary Incontinence
Brief Title: The Efficacy and Safety of Fotona Smooth® Device for the Treatment of Stress Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cork University Hospital (Other)
Collaborators: Fotona d.o.o. (Industry)
Responsible Party: Principal Investigator, Barry O'Reilly, Professor, Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FOTONA-Incontilase
Record Dates: First submitted 2017-03-20; First posted 2017-04-04 (Actual); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fotona Dynamis Er:YAG Laser System (Active Comparator): Active treatment with Fotona Dynamis Er:YAG Laser System
  Interventions: Device: Fotona Dynamis Er:YAG Laser System
- Fotona Dynamis Er:YAG Laser System with Sham handpience (Sham Comparator): Sham treatment with a sham handpiece and parameter presentations masked
  Interventions: Device: Fotona Dynamis Er:YAG Laser System with sham handpience

INTERVENTIONS:
Device: Fotona Dynamis Er:YAG Laser System — Treatment of urodynamic proven stress urinary incontinence using the Fotona Dynamis Er:YAG Laser System in the active arm
  Arms: Fotona Dynamis Er:YAG Laser System
Device: Fotona Dynamis Er:YAG Laser System with sham handpience — Sham treatment with a sham handpiece and parameter presentations masked
  Arms: Fotona Dynamis Er:YAG Laser System with Sham handpience

SUMMARY:
There are many existing treatments of female stress urinary incontinence such as the use of adult absorbent pads and diapers, behavioral training, including bladder training, pelvic muscle exercises, biofeedback, urethral plugs, intravaginal prosthesis, electrical stimulation, periurethral injections, and reconstructive surgery. However, there is still a lack of effective minimally invasive treatment options that are independent of patient compliance.

One emerging approach of minimally invasive SUI therapy is pelvic floor reinforcement using laser therapy.

The primary objective of this post-marketing study is to confirm the effectiveness and safety of the FotonaSmooth® device in the treatment of stress urinary incontinence (SUI) in a large number of females using objective and subjective methods.

Patients with stress incontinence will be assigned to two groups, an active group, where the Fotona Dynamis Er:YAG Laser System will be used, and a sham group where a very low laser setting will be used, and parameter presentations will be masked.

Participants will be adult females, 18 years old and older with clinical and urodynamic diagnosis of Stress Urinary Incontinence,who have had no significant improvement in urinary incontinence from at least one previous conservative treatment, such as behavioral measures, pelvic floor muscle training or the use of absorbent pads

DETAILED DESCRIPTION:
Prospective, randomized, 2-treatment, sham-controlled, single (patient only) blinded, study design using convenience sampling to enroll subjects as they present and are found to be eligible per the inclusion/exclusion criteria. This multicenter clinical trial utilizes a randomized assignment allocation schedule stratified by clinical site. Allocation rule pertains to the ratio of subjects in each treatment arm. Sampling rules pertain to the number of subjects in each active treatment arm.

Two treatment arms enrolled on a 2:1 ratio: Active arm is the Fotona Dynamis Er:YAG Laser System and the control arm is a sham treatment with a very low laser setting and parameter presentations masked. The active arm subjects will be followed out to 12 months post-treatment. The sham arm subjects will be followed out to 6 months and then offered the active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult Female, 18 years of age or older,
* Clinical and UDS diagnosis of Stress Urinary Incontinence,
* No significant improvement in urinary incontinence from at least one previous conservative treatments, such as behavioral measures, pelvic floor muscle training or the use of absorbent pads

Exclusion Criteria:

1. Pre-existing bladder pathology including prior radiation treatment
2. Pregnancy
3. BMI>35
4. Radical pelvic surgery or previous incontinence surgery
5. Urinary tract infection or other active infections of urinary tract or bladder
6. Endometriosis
7. Any form of pelvic organ prolapse greater than stage 2, according to POP-Q
8. Diagnosis of urge incontinence
9. Diagnosis of collagen disorders e.g. benign joint hypermobility / Elhers-Danlos / Marfans etc.
10. Incomplete bladder emptying
11. Vesicovaginal fistula
12. Fecal incontinence
13. Unwillingness or inability to complete follow-up schedule
14. Unwillingness or inability to give Informed Consent
15. Failure to comply with diary requirements during extended baseline period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Reduction in 1-hour pad weight between active and sham groups | 6 months post-treatment
  Reduction in 1-hour pad weight at 6 months post-treatment in active group vs the sham treated group at 6 months post treatment
Safety: Incidence and severity of device related Adverse Events | 6 months post-treatment
  Incidence and severity of device related Adverse Events (i.e., infections, edema, superficial burns, increased vaginal discharge, de novo urge incontinence).

SECONDARY OUTCOMES:
Durability of the effect | 12 months post-treatment
  Reduction in 1hr pad test weight in the treated group at 12 month follow-up vs. pad weight in the same group at baseline
Improvement | 6 and 12 months post-treatment
  Change in mean Cough Stress test score at 6 and 12 months post-treatment
Change in King's Health Questionnaire (KHQ) | from baseline to 6 and 12 months post-treatment.
  Change in mean KHQ from baseline to 6 and 12 months post-treatment
Change in mean PISQ-12 test scores | from baseline to 6 and 12 months post-treatment.
  Change in mean PISQ-12 test scores from baseline to 6 and 12 months post-treatment.
Subjective assessment of pain | 6 months
  Patient reported assessment of pain during treatment
Change in International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) score | from baseline to 6 and 12 months post-treatment.
  Change in mean ICIQ-SF from baseline to 6 and 12 months post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Barry O'Reilly, Professor, Principal Investigator — University College Cork
Locations (9):
- Lutheran Hospital Hagen-Haspe, Hagen, Germany
- University of Athens, Alexandra Hospital, Athens, Greece
- Cork Womens Clinic, Cork, Ireland
- University Clinical Centre, Ljubljana, Slovenia
- Switzerland (2):
  - Inselspital Bern, University Hospital, Bern
  - Cantonal Hospital Frauenfeld, Frauenfeld
- United Kingdom (3):
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Birmingham Women's Hospital NHS foundation trust, Birmingham
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ippolito GM, Crescenze IM, Sitto H, Palanjian RR, Raza D, Barboglio Romo P, Wallace SA, Orozco Leal G, Clemens JQ, Dahm P, Gupta P. Vaginal lasers for treating stress urinary incontinence in women. Cochrane Database Syst Rev. 2025 Jul 25;7(7):CD013643. doi: 10.1002/14651858.CD013643.pub2. PMID 40709601